CLINICAL TRIAL: NCT06614127
Title: Continuous Intraoperative Glucose Monitoring: A Pilot Study
Brief Title: Continuous Glucose Monitoring: A Pilot Study
Status: Active, not recruiting | Type: Observational
Sponsor: Loma Linda University (Other)
Responsible Party: Principal Investigator, Melissa McCabe, Associate Professor, Anesthesiology, Loma Linda University
Other Study IDs: IRB 5230596
Record Dates: First submitted 2024-08-27; First posted 2024-09-26 (Actual); Last update posted 2025-08-05 (Actual); Status verified 2025-06

CONDITIONS: Anesthesia
Keywords: Continuous Glucose Monitoring; Electrocautery

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (2):
- Continuous glucose monitoring site: upper arm: Adult, non-cardiothoracic surgical patients with Dexcom G7® sensor placed in upper arm over the deltoid
  Interventions: Device: Dexcom G7® sensor placed in upper arm and positioned over deltoid
- Continuous glucose monitoring site: anterior thigh: Adult, non-cardiothoracic surgical patients with Dexcom G7® sensor placed on the anterior aspect of the thigh
  Interventions: Device: Dexcom G7® sensor placed in anterior thigh

INTERVENTIONS:
Device: Dexcom G7® sensor placed in upper arm and positioned over deltoid — For the "subjects with Dexcom G7® sensor placed in the upper arm and positioned over the deltoid" cohort, study personnel will place the Dexcom G7® sensor on the subjects' deltoid and the electrodispursive pad on the thigh.
  Groups: Continuous glucose monitoring site: upper arm
Device: Dexcom G7® sensor placed in anterior thigh — For the "subjects with Dexcom G7® sensor place in anterior thigh" cohort, study personnel will place the Dexcom G7® sensor in the anterior thighs and the electrodispursive pad will be placed on the opposite thigh.
  Groups: Continuous glucose monitoring site: anterior thigh

SUMMARY:
The purpose of this study is to evaluate connectivity of the FDA approved DexCom G7® continuous glucose monitor in the operating room. Continuous glucose monitors are applied to the skin and a thin sampling filament is inserted into the skin and measures blood sugar in the interstitial fluid. The DexCom G7® is used regularly outside of the operating room to monitor blood sugar, however the use of the device in the operating room environment has been limited by connectivity issues. This study will assess device connectivity at different monitoring sites.

DETAILED DESCRIPTION:
This feasibility pilot study will assess connectivity of the DexCom G7® continuous glucose monitoring device (CGM) in the operating room environment at different locations on the body. The investigators believe device connectivity is affected by use of electrocautery. The monitoring sites were selected to limit electromagnetic interference from electrocautery.

One cohort will have the CGM device placed on the deltoid and the electrodispersive pad placed on the thigh and the other cohort will have the CGM device placed on the thigh with the electrodispersive pad on the opposite thigh.

Study personnel will note when electrocautery is used throughout the surgery and observe if the DexCom G7® continues to maintain connectivity with the receiver and provides a glucose reading. Comparing the timing of electrocautery use with connectivity to the DexCom G7® receiver provides important insight to the relationship between electrocautery and device connectivity.

The CGM readings will solely be used for feasibility purposes for this study and not for determining interventions for the subjects.

ELIGIBILITY:
Inclusion Criteria:

* Adults age 18 and above able to consent for themselves
* Willingness and ability to participate in study procedures
* Surgery length estimated 3 hours or longer

Exclusion Criteria:

* Cardiothoracic surgical patients
* Plan for intraoperative radiologic imaging
* Patients on IV infusion of insulin prior to surgery
* Anemia with hemoglobin less than 7
* Patients on hydroxyurea
* Patients with known adhesive allergies
* Pregnant women

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult non-cardiothoracic surgical patients.
Sampling Method: Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2024-10-24 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Effect of DexCom G7® sensor position on receiver connectivity during and after electrocautery use. | Change between baseline at start of procedure and completion of procedure, up to 6 hours.
  Connectivity will be recorded continuously from start to finish of the procedure.
  The percentage of time the Dexcom G7® device remains connected during the subject's surgical case will be measured. The effect of electrocautery on CGM connectivity will be assessed by comparing the start and stop times in connectivity to the start and stop times of electrocautery. Connectivity time greater than 80% is considered highly effective. Connectivity time between 20% and 80% is considered effective. Connectivity time less than 20% is considered sub-optimal.

CONTACTS AND LOCATIONS:
Overall Officials: Richard L Applegate, MD, Study Chair — Loma Linda University
Locations (1):
- Loma Linda University Troesch Medical Center, Loma Linda, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Singh LG, Satyarengga M, Marcano I, Scott WH, Pinault LF, Feng Z, Sorkin JD, Umpierrez GE, Spanakis EK. Reducing Inpatient Hypoglycemia in the General Wards Using Real-time Continuous Glucose Monitoring: The Glucose Telemetry System, a Randomized Clinical Trial. Diabetes Care. 2020 Nov;43(11):2736-2743. doi: 10.2337/dc20-0840. Epub 2020 Aug 5. PMID 32759361
- [Background] Sweeney AT, Pena S, Sandeep J, Hernandez B, Chen Y, Breeze JL, Bulut A, Feghali K, Abdelrehim M, Abdelazeem M, Srivoleti P, Salvucci L, Cann SB, Norman C. Use of a Continuous Glucose Monitoring System in High-Risk Hospitalized Noncritically Ill Patients With Diabetes After Cardiac Surgery and During Their Transition of Care From the Intensive Care Unit During COVID-19: A Pilot Study. Endocr Pract. 2022 Jun;28(6):615-621. doi: 10.1016/j.eprac.2022.03.001. Epub 2022 Mar 8. PMID 35276324
- [Background] Espinoza J, Xu NY, Nguyen KT, Klonoff DC. The Need for Data Standards and Implementation Policies to Integrate CGM Data into the Electronic Health Record. J Diabetes Sci Technol. 2023 Mar;17(2):495-502. doi: 10.1177/19322968211058148. Epub 2021 Nov 20. PMID 34802286
- [Background] Avari P, Lumb A, Flanagan D, Rayman G, Misra S, Dhatariya K, Choudhary P. Continuous Glucose Monitoring Within Hospital: A Scoping Review and Summary of Guidelines From the Joint British Diabetes Societies for Inpatient Care. J Diabetes Sci Technol. 2023 May;17(3):611-624. doi: 10.1177/19322968221137338. Epub 2022 Nov 28. PMID 36444418
- [Background] Renard E, Cobelli C, Kovatchev BP. Closed loop developments to improve glucose control at home. Diabetes Res Clin Pract. 2013 Nov;102(2):79-85. doi: 10.1016/j.diabres.2013.09.009. Epub 2013 Sep 28. PMID 24128998
- [Background] Dumitrascu AG, Perry MF, Boone RJ, Guzman MP, Chirila RM, McNally AW, Colibaseanu DT, Meek SE, Ball CT, White LJ, Chindris AM. Continuous Glucose Monitoring for Patients with COVID-19 Pneumonia: Initial Experience at a Tertiary Care Center. Endocr Pract. 2023 Mar;29(3):155-161. doi: 10.1016/j.eprac.2022.12.012. Epub 2022 Dec 22. PMID 36566985
- [Background] Adamska O, Mamcarz A, Lapinski M, Radzimowski K, Stepinski P, Szymczak J, Swiercz M, Zarnovsky K, Maciag BM, Stolarczyk A. Continuous glycemia monitoring in perioperative period in patients undergoing total knee or hip arthroplasty: A protocol for a prospective observational study. Medicine (Baltimore). 2022 Oct 21;101(42):e31107. doi: 10.1097/MD.0000000000031193. PMID 36281192
- [Background] Spanakis EK, Urrutia A, Galindo RJ, Vellanki P, Migdal AL, Davis G, Fayfman M, Idrees T, Pasquel FJ, Coronado WZ, Albury B, Moreno E, Singh LG, Marcano I, Lizama S, Gothong C, Munir K, Chesney C, Maguire R, Scott WH, Perez-Guzman MC, Cardona S, Peng L, Umpierrez GE. Continuous Glucose Monitoring-Guided Insulin Administration in Hospitalized Patients With Diabetes: A Randomized Clinical Trial. Diabetes Care. 2022 Oct 1;45(10):2369-2375. doi: 10.2337/dc22-0716. PMID 35984478
- [Background] Faulds ER, Dungan KM, McNett M. Implementation of Continuous Glucose Monitoring in Critical Care: A Scoping Review. Curr Diab Rep. 2023 Jun;23(6):69-87. doi: 10.1007/s11892-023-01503-5. Epub 2023 Apr 13. PMID 37052790
- [Background] Boeder S, Kulasa K. Hospital care: improving outcomes in type 1 diabetes. Curr Opin Endocrinol Diabetes Obes. 2021 Feb 1;28(1):14-20. doi: 10.1097/MED.0000000000000601. PMID 33315629
- [Background] Jackson MA, Ahmann A, Shah VN. Type 2 Diabetes and the Use of Real-Time Continuous Glucose Monitoring. Diabetes Technol Ther. 2021 Mar;23(S1):S27-S34. doi: 10.1089/dia.2021.0007. PMID 33534631